CLINICAL TRIAL: NCT04869488
Title: An Open, Multi-center, Phase Ⅱ Clinical Study of Fluzoparib Combined With Apatinib or Fluzoparib in the Treatment of Metastatic Castration-resistant Prostate Cancer
Brief Title: A Trial of SHR3162 Combined With Apatinib Mesylate Tablets or SHR3162 Monotherapy in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR3162-Ⅱ-202
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — fluzoparib; enzalutamide; Abiraterone Acetate; Prednisone; apatinib

STUDY DESIGN:
Intervention Model Description: Fluzopali in combination with apatinib mesylate or fluzopali monotherapy with or without homologous recombinant repair-related gene mutations in metastatic castration-resistant prostate in subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluzoparib (Experimental)
  Interventions: Drug: Fluzoparib
- Enzalutamide OR abiraterone acetate With Prednisone Acetate Tablets (Active Comparator)
  Interventions: Drug: Enzalutamide OR abiraterone acetate With Prednisone Acetate Tablets
- Fluzoparib Combined With Apatinib (Experimental)
  Interventions: Drug: Fluzoparib Combined With Apatinib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib Orally twice daily（Cohort 1、Cohort 4）
  Arms: Fluzoparib
Drug: Enzalutamide OR abiraterone acetate With Prednisone Acetate Tablets — Enzalutamide OR abiraterone acetate Orally once daily（Cohort 1）
  Arms: Enzalutamide OR abiraterone acetate With Prednisone Acetate Tablets
Drug: Fluzoparib Combined With Apatinib — Fluzoparib Orally twice daily; Apatinib Orally once daily（Cohort 2、Cohort 3、Cohort 4）
  Arms: Fluzoparib Combined With Apatinib

SUMMARY:
Main research purpose: To evaluate the effectiveness of Fluzoparib combined with apatinib mesylate in the treatment of patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. Age ≥18 years old;
3. Pathologically diagnosed metastatic castration-resistant prostate adenocarcinoma;
4. It is confirmed by the central laboratory based on tumor tissue or ctDNA detection that it is accompanied by germline or system homologous recombination repair-related gene mutations (Cohorts 4) or not accompanied by homologous recombination repair-related gene mutations (Cohort 2);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
6. Has a life expectancy of ≥ 12 weeks.

Exclusion Criteria:

1. Past (within 5 years) or concurrently suffering from other malignant tumors, except for cured skin basal cell carcinoma;
2. Subjects have used PARP inhibitors in the past, including but not limited to olaparib, niraparib, and lukapanib; or have used apatinib in the past; or have received mitoxantrone and cyclophosphamide in the past Treatment with amide or platinum-containing chemotherapeutics;
3. Severe bone injury caused by tumor bone metastasis, pathological fractures or spinal cord compression in important parts that occurred within 6 months before being informed or is expected to occur in the near future;
4. The subject has cancerous meningitis, or untreated central nervous system metastasis;
5. Those who cannot swallow pills normally, or have abnormal gastrointestinal function, which may affect drug absorption by the researcher;
6. Subjects with congenital or acquired immune deficiencies (such as HIV infection), or active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA ≥500 IU/ml; hepatitis C reference: HCV antibody positive and HCV virus copy number> upper limit of normal );
7. According to the judgment of the investigator, the subject has other factors that may cause the study to be terminated halfway, such as other serious diseases (including mental illness) that require combined treatment, severe laboratory abnormalities, family or society, etc. Factors that will affect the safety of subjects or the collection of data and samples.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Comprehensive response rate | up to 2 years
  Comprehensive remission rate means the proportion of objective remission or PSA remission evaluated by the investigator based on the RECIST v1.1 standard and the PCWG3 standard

SECONDARY OUTCOMES:
Radiological progression-free survival (rPFS) | up to 2 years
  The time from randomisation until the date of objective radiological disease progression (by RECIST 1.1 and Prostate Cancer Working Group 3 (PGWG-3)) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from randomised therapy or received another anti-cancer therapy prior to progression.
Objective response rate (ORR) | At the time point of every 8 weeks，up to 2 years
  ORR is the percentage of patients with at least one visit response of Complete response (CR) or Partial response (PR), in their soft tissue disease assessed by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), in the absence of progression on bone scan assessed by Prostate Cancer Working Group 3 (PCWG3)).
PSA response rate | At the time point of every 4 weeks，up to 2 years
  PSA response rate was Defined as the proportion of subjects whose serum PSA level decreased by ≥50% from baseline after treatment.
Time to PSA progression (PSA-TTP) | At the time point of every 4 weeks，up to 2 years
  PSA-TTP was defined as the time from random (cohort 1 and 4) or first medication (cohort 2 and 3) to the first progression of PSA; PSA progression is determined according to the PCWG3 standard, and changes in PSA levels within the 12 weeks before treatment (that is, before C4D1) are not included in this Evaluation.
Overall Survival (OS) | At the time point of every 2 months，up to 2 years
  Number of Participants with Overall Survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided